CLINICAL TRIAL: NCT01356186
Title: Pilot Trial of Inpatient Cognitive Therapy for the Prevention of Suicide in Military Personnel With Acute Stress Disorder of Post Traumatic Stress Disorder
Brief Title: Pilot Trial of Inpatient Cognitive Therapy for the Prevention of Suicide in Military Personnel
Acronym: CDMRP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Henry M. Jackson Foundation for the Advancement of Military Medicine (Other)
Collaborators: Congressionally Directed Medical Research Programs (U.S. Federal Agency)
Responsible Party: Principal Investigator, Marjan Holloway, Associate Professor, Henry M. Jackson Foundation for the Advancement of Military Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: W81XWH-08-2-1072
Record Dates: First submitted 2011-05-17; First posted 2011-05-19 (Estimated); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Suicide, Attempted
Keywords: Suicide; Cognitive Therapy; Inpatient; Military
MeSH Terms: conditions — Suicide, Attempted; Suicide | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Post Admission Cognitive Therapy (PACT) (Experimental): Six (6) 60-90 Minutes Sessions of Post Admission Cognitive Therapy Delivered Preferably Over 3 Consecutive Days of Inpatient Stay
  Interventions: Behavioral: Post Admission Cognitive Therapy (PACT)
- Enhanced Usual Care (EUC) (No Intervention): Treatment As Usual and Study Assessment Services

INTERVENTIONS:
Behavioral: Post Admission Cognitive Therapy (PACT) — Individual psychotherapy; 6 sessions; 60-90 minutes in duration; administered over preferably 3 days of psychiatric hospitalization
  Other Names: Cognitive Therapy; Cognitive Behavior Therapy
  Arms: Post Admission Cognitive Therapy (PACT)

SUMMARY:
The broad objective of this research is to effectively utilize a unique window of opportunity during the hospitalization period following a recent suicide attempt to deliver a brief and targeted intervention for traumatized individuals.

DETAILED DESCRIPTION:
Participation in military operations, especially in times of war, places personnel and their family members at increased risk for mental health problems. In 2003, among the 1.4 million active duty United States service members, mental disorders remained the leading cause of hospitalization for men and the second leading cause of hospitalization for women. Posttraumatic stress disorder (PTSD) and suicide behavior among military personnel are the leading causes of psychiatric hospitalization. Both are considered significant public health problems. Existing literature provides strong support for the relationship between PTSD and suicide ideation, attempts, and deaths. PTSD, in fact, shows the strongest association with suicide behavior of any of the anxiety disorders and has equal or greater odds ratio than mood disorders for resulting in impulsive suicide attempts. However, to date, no evidence-based interventions have been developed for individuals with PTSD who attempt suicide. Therefore, the investigators aim to develop, implement, and evaluate an inpatient based cognitive behavioral care plan for service members and beneficiaries, with symptoms of either Acute Stress Disorder (ASD) or PTSD, who are admitted for hospitalization following a recent suicide attempt.

The investigators will randomize 50 traumatized patients hospitalized at the Walter Reed Army Medical Center for a recent suicide attempt to one of two conditions: (1) Post-Admission Cognitive Therapy + Enhanced Usual Care (PACT+EUC) or (2) Enhanced Usual Care (EUC). Individuals who are over the age of 18, able to communicate in English and willing to provide informed consent will be recruited. The PACT+EUC condition will consist of six 1-hr individual cognitive therapy sessions administered over 3 days over the course of the patient's hospital stay. The EUC condition will consist of the usual care patients receive at an inpatient facility during their hospitalization in addition to assessment services provided by independent evaluators who work directly with our research team. The primary outcome variable is the number of subsequent suicide attempts. The investigators expect that patients in the control condition will reattempt suicide at an earlier date and at a higher frequency as compared to patients enrolled in the intervention condition. Secondary outcome measures include the severity of depression, hopelessness, suicide ideation, and post traumatic symptoms. Patients in both conditions will be assessed on the dependent measures at baseline and at 1-, 2-, and 3- month follow-up intervals. Data analyses will provide estimates of the level of improvement demonstrated by the intervention condition, PACT relative to the control condition, EUC over time.

The development and subsequent dissemination of innovative inpatient focused interventions for traumatized individuals with suicide attempt behavior will significantly contribute to our national and military suicide prevention objectives. The research aims to effectively utilize a unique window of opportunity during the hospitalization period following a recent suicide attempt to deliver a brief and targeted intervention to military personnel and family members diagnosed with a trauma-related condition. If our designed intervention demonstrates to be clinically feasible, acceptable, and associated with preliminary evidence of improvement in symptoms relative to the control condition, a larger randomized controlled trial will be proposed to definitively determine the efficacy of the intervention. Without adequate treatment, PTSD and suicide behavior may result in costly utilization of social services, human suffering, and eventual death. The Department of Veterans Affairs reports that veterans as compared to the general US population are at greater risk for suicide by almost 23%. The study targets at-risk individuals immediately following psychiatric hospitalization to minimize the likelihood of future complications as seen previously with Vietnam veterans. The projected time to achieve a consumer-related outcome would be 3-5 years.

ELIGIBILITY:
Inclusion Criteria

1. Suicide Attempt (Recent or Lifetime) Psychiatric Admission
2. History of Trauma
3. Baseline Completed within 48 Hours of Admission
4. Over the Age of 18
5. Provides Informed Consent

Exclusion Criteria

1. Self-Inflicted Harm with No Intent or Desire to Die
2. Medical Incapacity to Participate
3. Current State of Active Psychosis
4. Expected Discharge within 72 Hours of Admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2008-07; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Repeat Suicide Attempts | 1, 2, and 3 months
  The Columbia Suicide Severity Rating Scale (C-SSRS) will be used to assess for subsequent suicide attempts.

SECONDARY OUTCOMES:
Depression | 1, 2, and 3 months
  Depressive symptoms will be measured using the Beck Depression Inventory-II (BDI-II).
Hopelessness | 1, 2, and 3 months
  Levels of hopelessness will be assessed using the Beck Hopelessness Scale (BHS).
Suicide Ideation | 1, 2, and 3 months
  The Scale for Suicide Ideation (SSI) will be used to assess for suicide-related thoughts (ideations), as well as intensity, frequency, and specificity of any such thoughts.
Post-Traumatic Stress Symptoms | 1, 2, and 3 months
  The Clinician Assessments of PTSD Scale (CAPS) and the PTSD Checklist (PCL) will be used to assess for post-traumatic stress symptoms.
Reliable Change Index | 1, 2, and 3 months
  This is a statistical strategy to examine meaningful clinical change over time for one participant at a time.

CONTACTS AND LOCATIONS:
Overall Officials: Marjan Holloway, Ph.D., Principal Investigator — Uniformed Services University of the Health Sciences
Locations (2):
- United States (2):
  - Uniformed Services University of the Health Sciences, Bethesda, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ghahramanlou-Holloway M, Cox D, & Greene F. Post-admission cognitive therapy: A brief intervention for psychiatric inpatients admitted after a suicide attempt. Cognitive and Behavioral Practice 19: 233-244, 2012.
- [Background] Neely L, Irwin K, Carreno Ponce JT, Perera K, Grammer G, & Ghahramanlou-Holloway M. Post Admission Cognitive Therapy (PACT) for the prevention of suicide in military personnel with histories of trauma: Treatment development and case example. Clinical Case Studies, 12(6), 457-473, 2013.
- [Result] LaCroix JM, Perera KU, Neely LL, Grammer G, Weaver J, Ghahramanlou-Holloway M. Pilot trial of post-admission cognitive therapy: Inpatient program for suicide prevention. Psychol Serv. 2018 Aug;15(3):279-288. doi: 10.1037/ser0000224. PMID 30080085
- [Derived] Witt KG, Hetrick SE, Rajaram G, Hazell P, Taylor Salisbury TL, Townsend E, Hawton K. Psychosocial interventions for self-harm in adults. Cochrane Database Syst Rev. 2021 Apr 22;4(4):CD013668. doi: 10.1002/14651858.CD013668.pub2. PMID 33884617
- [Derived] LaCroix JM, Colborn VA, Hassen HO, Perera KU, Weaver J, Soumoff A, Novak LA, Ghahramanlou-Holloway M. Intimate partner relationship stress and suicidality in a psychiatrically hospitalized military sample. Compr Psychiatry. 2018 Jul;84:106-111. doi: 10.1016/j.comppsych.2018.04.006. Epub 2018 Apr 21. PMID 29747068